CLINICAL TRIAL: NCT02743273
Title: Identification of Prognostic Urinary Biomarker for Acute Kidney Injury in Preterm Infants by Proteomics
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Director of Neonatal Intensive Care Unit, Seoul National University Hospital
Other Study IDs: 1507-028-686
Record Dates: First submitted 2015-12-09; First posted 2016-04-19 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical definitions of acute kidney injury (AKI) have been based on an increase in serum creatinine and a decrease in urine output. However, applying this definition to neonates remains challenging because of the normal renal physiologic features that serum creatinine levels are expected to increase in the first days after birth, and impaired sodium reabsorption and concentrating ability.

Because of several limitations of early detection of AKI, investigators are focused on identifying biomarkers that predict AKI before an increase serum creatinine level.

Investigators will collect urine from preterm infants before and after administrating ibuprofen for closing patent ductus arteriosus. To identify novel biomarkers, investigators will analyze urine by proteomics. To verify those biomarkers, investigators will use initial urine on the first day of life from preterm infants who diagnosed AKI within 7 days after birth without any risk factors for AKI and enrolled institutional bio-repository.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 32 weeks gestational age or birth weight less than 1,500 g admitted to the neonatal intensive care unit at Seoul National University Children's hospital

Exclusion Criteria:

* Congenital heart disease
* Known major congenital anomalies of the kidney and urinary tract
* Other genetic syndromes or medical conditions that preclude enrollment per judgement of the attending neonatologist

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Preterm infants with gestational age<32 weeks or birth weight<1,500 g who enrolled our institutional prospective cohort study for biorepository.
  2. Preterm infants with gestational age<32 weeks or birth weight< 1,500 g who need ibuprofen treatment for closing patent ductus arteriosus.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
change the level of novel urinary biomarkers after ibuprofen administration | change from 1 day before ibuprofen administration to 1 day after ibuprofen administration

SECONDARY OUTCOMES:
The level of novel urinary biomarkers in initial urine | within 24 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD., Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes